CLINICAL TRIAL: NCT05260060
Title: Youth Metacognitive Therapy (YoMETA): A Single-Blind Parallel Randomised Feasibility Trial
Brief Title: Youth Metacognitive Therapy Feasibility Trial
Acronym: YoMETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Greater Manchester Mental Health NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Adrian Wells, Professor of Clinical and Experimental Psychopathology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS ID: 296079
Record Dates: First submitted 2022-02-07; First posted 2022-03-02 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Child Mental Disorder; Anxiety Disorders; Depression
Keywords: Metacognitive Therapy; Feasibility; Anxiety; Depression; Mental health
MeSH Terms: conditions — Neurodevelopmental Disorders; Anxiety Disorders; Depression; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Chief investigator, research assistants and statisticians will be blind to treatment allocation of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Treatment (Control) (Active Comparator): Participants allocated to the control group will receive treatment as usual under the child and adolescent mental health service.
  Interventions: Behavioral: Treatment as usual: Control
- Group MCT (Intervention) (Experimental): Participants allocated to the intervention group will receive group metacognitive therapy sessions.
  Interventions: Behavioral: Group Metacognitive Therapy (Group-MCT): Experimental

INTERVENTIONS:
Behavioral: Treatment as usual: Control — Treatment usually delivered in service that may include but is not limited to cognitive behaviour therapy, exposure, eye movement desensitisation and reprocessing , behaviour therapy, family therapy.
  Arms: Usual Treatment (Control)
Behavioral: Group Metacognitive Therapy (Group-MCT): Experimental — Group metacognitive therapy (Group-MCT) focuses on developing adaptive control of worry, repetitive negative thinking and attention and modifies beliefs that maintain unhelpful thinking patterns. Treatment is 6 to 8 weekly sessions delivered by two trained mental health professionals, guided by a treatment manual, lasting approximately 90 minutes each session.
  Arms: Group MCT (Intervention)

SUMMARY:
One in eight children and young people (CYP) suffer mental health problems needing support or treatment and 5% have more than one such problem. The effects can be major, affecting CYP emotionally and functionally, impacting progress at school, relationships with others and increasing long term risk of mental health problems. Parents, schools, policy makers and the NHS often struggle to find the best way to help, especially within their limited budgets. The UK Government and the NHS have highlighted the need to improve mental health in CYP.

The most common treatment is cognitive behavioural therapy; however this can be time consuming, needs to be delivered over many weeks, must focus on the most upsetting problem first and is not very effective. One way to overcome this is to evaluate a group therapy that can treat multiple mental health problems at once. This new treatment is called Metacognitive Therapy (MCT).

The aim of the study is to see if participating in a randomized trial of Group MCT is a feasible and acceptable treatment for CYP suffering with anxiety, stress, depression, or a combination in comparison to usual care. This allows us to test key questions about recruitment and drop-out rates, test the protocol, and gain information about MCT including training and supervision needs of clinicians and the experience of patients receiving it.

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment for emotional disorder symptoms (i.e. generalized anxiety disorder, panic disorder, agoraphobia, post-traumatic stress disorder, obsessive compulsive disorder, social anxiety and/or depression).
* Native fluency in English language
* Medication permitted but must be stabilised for 6 weeks.

Exclusion Criteria:

* Presence of significant risk or safeguarding concerns
* Head injury/organic impairment
* Formal diagnosis or under assessment for Autism Spectrum Disorder or Attention Deficit-Hyperactivity Disorder
* Eating Disorder

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Revised Children Anxiety and Depression Scale - Short Version (RCADS) | Baseline, 20 weeks follow up, 32 weeks follow up, 44 weeks follow up
  Youth self-report questionnaire measuring total anxiety, total depression and total anxiety and depression.
  This is a feasibility study and therefore it is not primarily powered to detect a difference (change in scores). The principal aim is to test the feasibility of a study using. Here we are testing the feasibility of using the measures (RCADS), therefore the measures will be assessed by monitoring descriptive data and the analysis of complete data once follow up has been completed. Specifically, range in scores, number of complete measures, proportion of missing data. Analyses of outcomes (change) will focus on descriptive statistics and confidence intervals for treatment effects.

SECONDARY OUTCOMES:
Strength and Difficulties Questionnaire (SDQ) | Baseline, 20 weeks follow up, 32 weeks follow up, 44 weeks follow up
  Measure of psychological well-being across five subscales: emotion, hyperactivity, conduct, peer relations and pro-social behaviour.
  Feasibility of the measure will be assessed by monitoring descriptive data and the analysis of complete data once follow up has been completed. Analyses of outcomes (change) will focus on descriptive statistics and confidence intervals for treatment.
Metacognition Questionnaire - Adolescent Version (MCQ-A) | Baseline, 20 weeks follow up, 32 weeks follow up, 44 weeks follow up
  Measure of metacognitive beliefs across five subscales: positive beliefs about worry, negative beliefs about uncontrollability and danger, cognitive confidence, cognitive self-consciousness and cognitive control.
  Feasibility of the measure will be assessed by monitoring descriptive data and the analysis of complete data once follow up has been completed. Analyses of outcomes (change) will focus on descriptive statistics and confidence intervals for treatment.
Mood & Feelings Questionnaire (MFQ) | Baseline, 20 weeks follow up, 32 weeks follow up, 44 weeks follow up
  Measure of depressive symptoms in 6-17 year olds.
  Feasibility of the measure will be assessed by monitoring descriptive data and the analysis of complete data once follow up has been completed. Analyses of outcomes (change) will focus on descriptive statistics and confidence intervals for treatment.
Child Health Utility - 9D (CHU-9D) | Baseline, 20 weeks follow up, 32 weeks follow up, 44 weeks follow up
  Measure of paediatric quality of life using dimensions: worried, sad, pain, tired, annoyed, school/homework, sleep, daily routine, ability to join in activities.
  Feasibility of the measure will be assessed by monitoring descriptive data and the analysis of complete data once follow up has been completed. Analyses of outcomes (change) will focus on descriptive statistics and confidence intervals for treatment.
Health and Social Case Service-Use Interview (SUI) | Baseline, 20 weeks follow up, 32 weeks follow up, 44 weeks follow up
  Assessment of the child's use of primary, secondary or community-based health and social care services and how often they have used the service in the last 16 weeks or since last study assessment.

OTHER OUTCOMES:
Other Feasibility Outcomes | Baseline, 20 weeks follow up, 32 weeks follow up, 44 weeks follow up
  Feasibility will also be assessed using referral rates (Baseline), recruitment and retention rates (Baseline, 20 week, 32 weeks and 44 weeks), participant attendance at treatment sessions, and willingness to be randomized to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Wells, Principal Investigator — University of Manchester
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Derived] Wells A, Carter K, Hann M, Shields G, Wallis P, Cooper B, Capobianco L. Youth Metacognitive Therapy (YoMeta): protocol for a single-blind randomised feasibility trial of a transdiagnostic intervention versus treatment as usual in 11-16-year-olds with common mental health problems. Pilot Feasibility Stud. 2022 Sep 12;8(1):207. doi: 10.1186/s40814-022-01162-5. PMID 36096940
- See also: Research Project Website Page — https://adept-ru.com/research-projects/yometa/